CLINICAL TRIAL: NCT03092687
Title: Procedures for Sample Acquisition and Distribution for The Human Brain Collection Core
Status: Terminated | Type: Observational
Why Stopped: Not considered to be human subjects research
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917073; 17-M-N073
Record Dates: First submitted 2017-03-23; First posted 2017-03-28 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia; Major Depression; Bipolar Disorder; PTSD
Keywords: Mental Illness; Aging; Normal Development
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Bipolar Disorder; Stress Disorders, Post-Traumatic; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- psychiatric disorders: decedents with and without psychiatric use disorders
- substance disorders: decedents with and without substance use disorders

SUMMARY:
Background:

The Human Brain Collection Core (HBCC) collects brain and other tissues. They get these from deceased people who may or may not have had psychiatric disorders. The next of kin gives permission for researchers to get the tissues. Researchers want to collect medical details of people whose brains are donated. They also want to use the donated tissue to study brain chemistry and structure. This could lead to better treatments for mental illness.

Objective:

To create a collection of human brain tissue to learn about the causes and mechanisms of mental disorders.

Eligibility:

People willing to donate their deceased relative s brain tissue. The deceased person could not have had any of the following:

Severe mental retardation

Long-lasting seizure disorder

Infections that affect the brain

Decomposition

Brain damage

Being on a respirator for more than 12 hours

Major sepsis

Serious renal or hepatic disease

Certain dementias and degenerative diseases

Design:

Medical Examiner s Offices will screen donors who have recently died. Some others will be screened by hospitals or funeral homes.

Participants will be the next of kin. They will give consent for HBCC to obtain brain tissue from the deceased person. The tissue will be frozen for future research.

Participants will have a 30-minute phone call. They will answer questions about the deceased person s medical and psychiatric conditions. They will answer questions about the person s use of medicines and drugs.

Participants will be contacted by a social worker. They will be asked for permission to access the deceased person s medical records.

DETAILED DESCRIPTION:
Objective: The mission of Human Brain Collection Core (HBCC) is to gain insight into the causes and mechanisms of mental disorders.

Study Population: To be able to conduct this research, we obtain brain and other tissues from deceased individuals with and without psychiatric disorders.

Study Design: This protocol provides the ethical and scientific framework for tissue donations through referrals from Offices of the Chief Medical Examiners, hospitals or funeral homes. The next of kin are contacted to give permission for brain donation from the deceased. Once the tissue is obtained, it is frozen, catalogued and processed for distribution to other researchers and for in-house analysis. The HBCC dissects specific brain tissues based on request. All collaborations are subject to approval by an oversight committee. Currently, HBCC can leverage over 1,000 brains from a variety of psychiatric disorders and non-psychiatric subjects.

Outcome measures: Outcomes vary with specific collaborations, but include characterization of DNA, RNA, protein and other brain constituents that provide unique information at the molecular level. The data thus obtained are expected to provide new insights into brain physiology and the molecular pathology of psychiatric disorders, possibly leading to the identification of new therapeutic targets.

ELIGIBILITY:
* INCLUSION CRITERIA:

Brain tissue is needed from individuals suffering from a variety of neuropsychiatric disorders, including schizophrenia, anxiety disorders, suicide, bipolar disorder, depression, and substance use disorders (cocaine, alcohol, heroin or the like). In addition, brains from individuals without a history of neuropsychiatric disease will be needed as controls.

EXCLUSION CRITERIA:

An assessment is carried out on the information available from the referral source (generally a Medical Examiner s Office) prior to obtaining consent. This information is usually very succinct, indicating how the decedent was found and, if known, whether they had some psychiatric or obvious medical history. The following cases will be

excluded from collection:

* Severe mental retardation.
* Well documented, long lasting seizure disorder.
* Infections known to affect the brain such as syphilis, tuberculosis, with the exception of HIV infection.
* The body is decomposed. We consider collecting the brain up to three days after death.
* There is obvious damage to the brain by closed head injury or other trauma (gunshot wound, fall, etc.).
* There are brain infarcts, hemorrhages, tumors, stroke, or other brain lesions that destroy the normal brain structure.
* The patient has been maintained on a respirator (ventilator) for more than 12 hours in the period immediately prior to death.
* Major sepsis.
* Serious renal or hepatic disease.
* Multiple sclerosis (MS), Alzheimer s disease and other dementias and degenerative diseases.
* Known infection with Hepatitis C

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community Samples
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
To accumulate a vast repository of human brain tissues and characterize molecular signatures of psychiatric disorders using techniques such as genome-wide association analyses, DNA methylation, acetylation and chromatin modification patterns, RN... | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Marenco, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States